CLINICAL TRIAL: NCT00770718
Title: A Comparison of Recombinant Activated Factor VII, Prothrombin Complex Concentrate, and Fresh Frozen Plasma for Anticoagulation Reversal in Warfarin-Associated Acute Intracranial Hemorrhage: A Dose Ranging Pilot Study
Brief Title: Factor VII, Prothrombin Complex Concentrate, and Fresh Frozen Plasma in Warfarin-Related Intracranial Hemorrhage
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: University of Utah (Other)
Collaborators: Sheila B. Terry Memorial Research Fund (Other)
Responsible Party: Bradley Duhon, M.D./Resident, Department of Neurosurgery, University of Utah Department of Neurosurgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21152
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Intracranial Hemorrhage
Keywords: intracranial hemorrhage; warfarin; anticoagulant; Factor VII; Prothrombin
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — recombinant FVIIa; Factor IX; Profilnine SD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Recombinant Activated Factor VII (Experimental): The first five patients who meet the selection criteria will be administered an intravenous dose of rFVIIa 1mg upon arrival. INR will be drawn at 20 minutes post-rFVIIa administration. If normalized (≤1.3), then repeat INR with be drawn every 2 hours thereafter for 6 hours total, and again at 24 hours after initial administration. If at any time, the INR is >1.3, then rFVIIa 1mg will be readministered and the INR will again be checked 20 minutes after administration and every 2 hours for 6 hours total and again at 24 hours post-administration. This may be repeated until a total dose of 80mcg/kg has been given. If a maximum total of 80mcg/kg has been administered without successful correction of INR, then FFP infusions will be utilized to complete correction.
  Interventions: Drug: Recombinant Activated Factor VII (rFVIIa)
- Prothrombin Complex Concentrate (PCC) (Experimental): 5 patients will receive PCC based on ideal body weight. Each patient will receive 30 i.u./kg ideal body weight as is rounded to the nearest dispensed vial size. Vials are dispensed as 5mL (500 i.u.), 10mL (1000 i.u.), or 10mL (1500i.u.). INR will be drawn at 20 minutes post-administration and, if normalized (≤1.3), 2 hours post-administration and every 2 hours for 6 hours total. The INR will also be checked 24 hours post-administration. If at any time, the INR is >1.3, then PCC will be readministered at the same dose and the INR will again be checked 20 minutes after administration and every 2 hours for 6 hours total and again at 24 hours post-administration. A maximum total of 60 iu/kg can be administered before FFP will be used to complete the correction.
  Interventions: Drug: Prothrombin Complex Concentrate
- Fresh Frozen Plasma (FFP) (Active Comparator): The last five patients will receive transfusions of FFP to normalize INR. If the initial INR is between 2-4, then 2 units of FFP (Round 1) will be administered emergently. If the initial INR is >4, then 4 units of FFP will be administered (Round 1). The INR will be checked after each round of FFP infusion completed. Once INR ≤1.3, then the INR will be again checked every 2 hours after normalization for 6 hours total and then 24 hours post-initial infusion. If the INR should ever return to >1.3, then repeat infusions of FFP will begin as outlined above and the INR will be checked serially as defined above.
  Interventions: Biological: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Recombinant Activated Factor VII (rFVIIa) — Five patients who meet the selection criteria will be administered an intravenous dose of rFVIIa 1mg upon arrival. INR will be drawn at 20 minutes post-rFVIIa administration. If normalized (≤1.3), then repeat INR with be drawn every 2 hours thereafter for 6 hours total, and again at 24 hours after initial administration. If at any time, the INR is >1.3, then rFVIIa 1mg will be readministered and the INR will again be checked 20 minutes after administration and every 2 hours for 6 hours total and again at 24 hours post-administration. This may be repeated until a total dose of 80mcg/kg has been given.
  Other Names: Novoseven®
  Arms: Recombinant Activated Factor VII
Drug: Prothrombin Complex Concentrate — 5 patients will receive PCC based on ideal body weight. Each patient will receive 30 i.u./kg ideal body weight as is rounded to the nearest dispensed vial size. Vials are dispensed as 5mL (500 i.u.), 10mL (1000 i.u.), or 10mL (1500i.u.). INR will be drawn at 20 minutes post-administration and, if normalized (≤1.3), 2 hours post-administration and every 2 hours for 6 hours total. The INR will also be checked 24 hours post-administration. If at any time, the INR is >1.3, then PCC will be readministered at the same dose and the INR will again be checked 20 minutes after administration and every 2 hours for 6 hours total and again at 24 hours post-administration. A maximum total of 60 iu/kg can be administered.
  Other Names: Profilnine®
  Arms: Prothrombin Complex Concentrate (PCC)
Biological: Fresh Frozen Plasma — Five patients will receive transfusions of FFP to normalize INR. If the initial INR is between 2-4, then 2 units of FFP (Round 1) will be administered emergently. If the initial INR is >4, then 4 units of FFP will be administered (Round 1). The INR will be checked after each round of FFP infusion completed. Once INR ≤1.3, then the INR will be again checked every 2 hours after normalization for 6 hours total and then 24 hours post-initial infusion. If the INR should ever return to >1.3, then repeat infusions of FFP will begin as outlined above and the INR will be checked serially as defined above.
  Other Names: FFP
  Arms: Fresh Frozen Plasma (FFP)

SUMMARY:
The purpose of this dose-ranging pilot study is to compare Recombinant Activated Factor VII, Prothrombin Complex Concentrate and Fresh Frozen Plasma (each starting at low doses with escalation if necessary) for the reversal of warfarin in the setting of acute intracranial hemorrhage.

DETAILED DESCRIPTION:
Both recombinant activated Factor VIIa (rFVIIa) as well as Prothrombin Complex Concentrate (PCC) are labeled for the treatment of bleeding episodes in patients with hemophilia. Many hospitals are also using each for the following unlabeled indications: bleeding rescue in surgical patients, severe multiple trauma with ongoing bleeding, intracranial bleeding < 4 hours since symptom onset, traumatic head injury with evidence of expanding bleed, retroperitoneal bleed, and life-threatening bleeding due to idiopathic coagulopathy. To our knowledge, these two products have never been clinically compared head to head for the reversal of warfarin in the setting of intracranial hemorrhage.

The rFVIIa (Novoseven) guidelines are based off of national data and utilize a dose range of 40-90 mcg/kg of ideal body weight (2.8-6.3 mg for a 70 kg. patient) with an additional dose if needed. The dose cited in the literature for the management of intracerebral bleeds ranges from 10 to 120 mcg/kg (0.7 - 8.4 mg for a 70 kg. patient,) with higher doses associated with increased risk of thromboembolic events.

The recommended dosing of PCC is 30-50 i.u. per kilogram of ideal body weight with additional dosing if needed. PCC (Profilnine®SD) is a mixture of the following vitamin K-dependent clotting factors: II (prothrombin), VII (proconvertin), IX (plasma thromboplastin component; PTC; Christmas factor), and X (Stuart-Prower factor). These factors are required for the conversion of prothrombin to thrombin and thus adequate hemostasis, and are synthesized in the liver.

Currently at the most hospitals around the country, fresh frozen plasma (FFP) is the mainstay for reversal of warfarin-related coagulopathy in intracranial hemorrhage at the discretion of the treating attending physician. We propose to study all the current reversal practices in the intracranial hemorrhage population here at the University of Utah as part of a quality improvement project for both patient safety and cost.

We will perform a safety and feasibility study comparing dosage regimens of rFVIIa, FIXa and fresh frozen plasma (FFP) infusion in the normalization of coagulopathy in the context of warfarin-related intracerebral hemorrhage. Our primary outcome is time to INR normalization defined as INR≤ 1.3 on two consecutive readings separated by 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic intracranial hemorrhage (subdural or intraparenchymal)
* Known warfarin ingestion
* INR ≥2.0
* GCS <13

Exclusion Criteria:

* Pregnancy
* History of venous thrombosis or pulmonary embolus
* Acute myocardial infarction
* Acute stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Normalization of INR (<1.4) | 20min, 2hrs, 4hrs, 6hrs, 24hrs

SECONDARY OUTCOMES:
Hematoma progression | 24hrs
Neurological status | 24hrs & 1month
Timing of intervention completion | 24hrs
Dosing of intervention required | 24hrs
Medical complications during hospitalization | days